CLINICAL TRIAL: NCT05544890
Title: Core Stability (Therapeutic) Exercise Alone or in Combination With Manual Therapy or Kinesio Tape in Patients With Chronic Low Back Pain: Randomized Control Trial.
Brief Title: Effects of Core Exercise in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCV/2019-2020/138
Record Dates: First submitted 2022-09-08; First posted 2022-09-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Low Back Pain
Keywords: Chronic pain; Muskuloskeletal manipulation; Complementary therapies; Catastrophization; Kinesiophobia
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Kinesiophobia | interventions — Exercise; Musculoskeletal Manipulations; Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The groups will be arranged randomly and the masking technique to be used will be the doble blind procedure. The subjects will be randomly selected through the EPIDAT 4.2 program. The random allocation to each group will be made just by one external researcher, this way, neither the main researcher, nor the participants, will know their allocation. Furthermore, the inspector who will collect the evaluation data won´t know the allocation of each subject.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapeutic exercise Group (ET) (Active Comparator): The ET group is going to follow a program of core stabilization through specific therapeutic exercise. Two weekly sessions will be programmed for 12 weeks, making a total of 24 sessions. Each session will have a duration of 60 minutes. All patients will start learning how to activate the transversus abdominal muscle in the first training session. The exercises will be made in 1 to 3 series of among 8 and 15 repetitions and the isometric contractions for 5 to 10 seconds. The rest between series will be of 30 seconds, and between exercise of 2-3 minutes.
  Interventions: Procedure: Exercise
- Manual Therapy group (ETmanualtherapy) (Active Comparator): Prior the core exercise previously exposed in group ET, group ETmanualtherapy will lay on the stretcher, where the physiotherapist will work on a manual therapy thrust. The participant will receive a high velocity and low range impulse technique in lateral position on both sides.
  Interventions: Procedure: Exercise; Procedure: Manual Therapy
- Kinesiotape Group (ETkinesiotape) (Active Comparator): The ETkinesiotape will go previously through physiotherapy, where a kinesiotape band will be applied (Kinesiotape "Nondolens" 5cmx5cm black color), in Y technique, by applying the kinesiotape base in neutral position of the lumbar spine without any tension on the tape. The participants realize the same exercise program than the other groups plus the kinesiotape applied.
  Interventions: Procedure: Exercise; Procedure: Kinesiotape

INTERVENTIONS:
Procedure: Exercise — All patients will start learning how to activate the transversus abdominal muscle in the first training session. The exercises will be made in 1 to 3 series of among 8 and 15 repetitions and the isometric contractions for 5 to 10 seconds. The rest between series will be of 30 seconds, and between exercise of 2-3 minutes.
  Other Names:
  - Therapeutic exercise
Procedure: Manual Therapy — All patients will start learning how to activate the transversus abdominal muscle in the first training session. The exercises will be made in 1 to 3 series of among 8 and 15 repetitions and the isometric contractions for 5 to 10 seconds. The rest between series will be of 30 seconds, and between exercise of 2-3 minutes.
  Other Names:
  - Manipulation
  Arms: Manual Therapy group (ETmanualtherapy)
Procedure: Kinesiotape — All patients will start learning how to activate the transversus abdominal muscle in the first training session. The exercises will be made in 1 to 3 series of among 8 and 15 repetitions and the isometric contractions for 5 to 10 seconds. The rest between series will be of 30 seconds, and between exercise of 2-3 minutes.
  Other Names:
  - Kinesiotaping
  Arms: Kinesiotape Group (ETkinesiotape)

SUMMARY:
Non-specific low back pain in one of the main causes of disability for health care worldwide. The effectiveness of therapeutic exercise, of kinesio tape and of manual therapy in the treatment of low back pain is evaluated, but not a comparison of these techniques. Moreover, can these techniques be combined?

DETAILED DESCRIPTION:
Non-specific low back pain is one of the main causes of disability for health care worldwide. Nowadays, the mostly used technique to research low back muscular activity in electromyography.

Among the published studies, the effectiveness of therapeutic exercise, of kinesio tape and of manual therapy in the treatment of low back pain is evaluated, but not a comparison of these techniques.

Therefore, the purpose of this study was to investigate the effects of core stability exercise alone or in combination with manual therapy or kinesiotape on pain, dysfunction, psychosocial factors and pressure pain threshold (PPTs) in patients with low back pain in ODI stage 2. The investigators hypothesized that exercise combined with manual therapy would provide greater changes and benefits than exercise alone.

This study's population will be composed by at least 15 individuals per group, both the male and female, with ages among 20 and 60.

Participants will be randomly and blindly divided in three groups of intervention. The three groups will be: Exercise group or ET (realize therapeutic exercise alone), manual therapy group o ETmanualtherapy (realize manual therapy prior therapeutic exercise), and kinesiotape group or ETkinesiotape (realize therapeutic exercise plus kinesiotape).

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of CLBP confirmed by an orthopaedic specialist Classification at Stage 2 by ODI Not receiving pharmacological treatment such as anti-inflammatories or corticosteroids.

Exclusion Criteria:

* Previous or scheduled surgeries in the low back and abdominal area
* Presence of severe fractures or pathologies.
* Diagnosis of radiculopathy or neuropathy (with or without spinal canal stenosis).
* Structural deformity in the spinal column.
* Neurological or psychiatric disorder.
* Presence or suspicion of pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index. | 12 weeks
  The Oswestry Disability Index (ODI) test will be made to all participants at three months. Divided into 10 sections (each is scored from zero to five, with higher scores meaning higher disability), it is self-administered to assess the limitations of different activities of daily living. That is why, it has been established that all participants in Stage 2 of the test are subsidiaries to make all the treatment modes of the study (manual therapy, kinesiotape and exercise). This way, we are able to rise the homogeneity that imposes a diagnostic label such as the chronic low back pain.

SECONDARY OUTCOMES:
Catastrophism (PCS) | 12 weeks
  To quantify the degree of catastrophism in the present study, the validated spanish version will be used as the pain catastrophism scale (PCS). The PCS is a 13-item self-report scale of 13 items, that presents same factor structure composed of the factors of rumination, despair and magnification. For each of these factors, it is given a value of 0 (without agreement) to 4 (always), so that at the end the examiner obtains a score between 0 and 52. Low scores indicate a low level of catastrophism and high values show high levels of catastrophism.
Kinesiophobia (TKS) | 12 weeks
  The mostly used questionnaire to evaluate kinesiophobia is the TKS (Tampa Kinesiophobia Scale) questionnaire, which we will use to measure which is the fear to movement of patients of low back pain. This scale includes work related lesions, lesions due to repetitive effort, relapses and the avoidance-fear. The questionnaire is composed of 17 items in which there is a differentiation between the negative and positive elements.
  This questionnaire will be filled in based on a Likert sale which ranges between 0 and 5, being 0 never and 5 always. The total punctuation ranges between 17 and 68, the higher the rate, the higher the degree of kinesiophobia.
Visual analog scale (VAS) | 12 weeks
  The VAS from 0 to 100, the scale considered to be the most representative, with the VAS being the best option due to its easy understanding and handling. This scale constitutes an effective tool to subjectively quantify this range, more discriminating than the scale that establishes its values from 0 to 10. This way, 0 will be considered as non-existent pain reflected by the individual and 10 as the worst pain imaginable by the patient.
Self-efficacy:questionnaire | 12 weeks
  To assess self-efficacy, it will be used the Chronic Pain Self-Efficacy Questionnaire, which assesses a person's belief in their ability to perform a specific behavior. It consists of 19 items, a Likert-type scale, and a response range of 0 to 10, where 0 is equivalent to feeling totally incapable, 5 moderately incapable and 10 fully capable. The result determines that the higher the score, the greater the degree of self-efficacy.
Pressure pain threshold | 12 weeks
  Pressure pain threshold (PPTs) is considered a useful method to calculate the degree of sensitization of deep tissues. It will be carried out using an algometer, which in this study will consist of a manometer attached to a cylindrical rubber tip. The manometer measures the pressure applied through the rubber and the patient should signal when this pressure starts being painful). Algometry is a widely studied and validated technique to quantify sensitivity in the diagnosis of symptomatic points and myofascial trigger points. The reliability of pressure pain threshold is relatively high, presenting coefficients of 0.9 and 0.95.
Electromyography | 12 weeks
  To obtain an objective measure of the muscle activation, surface electromyography will be used to evaluate the main core muscles - basically the rectus abdominis and multifidus.
  The electromyograph to be used will be the FREEEMG model of the brand BTS Bioengineering. It is a wireless electromyograph with probes attached to the prefilled electrodes, which collect the information. No additional hardware is required, as the same software processes the information taken. The data resolution is 16 bit and the frequency of 1 kHz.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Blanco, PDI, Principal Investigator — Doctoral School. Catholic University of Valencia San Vicente Mártir
Locations (1):
- Universitat Jaume I, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoy D, March L, Brooks P, Blyth F, Woolf A, Bain C, Williams G, Smith E, Vos T, Barendregt J, Murray C, Burstein R, Buchbinder R. The global burden of low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Jun;73(6):968-74. doi: 10.1136/annrheumdis-2013-204428. Epub 2014 Mar 24. PMID 24665116
- [Background] Finucane LM, Downie A, Mercer C, Greenhalgh SM, Boissonnault WG, Pool-Goudzwaard AL, Beneciuk JM, Leech RL, Selfe J. International Framework for Red Flags for Potential Serious Spinal Pathologies. J Orthop Sports Phys Ther. 2020 Jul;50(7):350-372. doi: 10.2519/jospt.2020.9971. Epub 2020 May 21. PMID 32438853
- [Background] Pitcher MH, Von Korff M, Bushnell MC, Porter L. Prevalence and Profile of High-Impact Chronic Pain in the United States. J Pain. 2019 Feb;20(2):146-160. doi: 10.1016/j.jpain.2018.07.006. Epub 2018 Aug 7. PMID 30096445
- [Background] Ketenci A, Zure M. Pharmacological and non-pharmacological treatment approaches to chronic lumbar back pain. Turk J Phys Med Rehabil. 2021 Mar 4;67(1):1-10. doi: 10.5606/tftrd.2021.8216. eCollection 2021 Mar. PMID 33948537
- [Background] Kreiner DS, Matz P, Bono CM, Cho CH, Easa JE, Ghiselli G, Ghogawala Z, Reitman CA, Resnick DK, Watters WC 3rd, Annaswamy TM, Baisden J, Bartynski WS, Bess S, Brewer RP, Cassidy RC, Cheng DS, Christie SD, Chutkan NB, Cohen BA, Dagenais S, Enix DE, Dougherty P, Golish SR, Gulur P, Hwang SW, Kilincer C, King JA, Lipson AC, Lisi AJ, Meagher RJ, O'Toole JE, Park P, Pekmezci M, Perry DR, Prasad R, Provenzano DA, Radcliff KE, Rahmathulla G, Reinsel TE, Rich RL Jr, Robbins DS, Rosolowski KA, Sembrano JN, Sharma AK, Stout AA, Taleghani CK, Tauzell RA, Trammell T, Vorobeychik Y, Yahiro AM. Guideline summary review: an evidence-based clinical guideline for the diagnosis and treatment of low back pain. Spine J. 2020 Jul;20(7):998-1024. doi: 10.1016/j.spinee.2020.04.006. Epub 2020 Apr 22. PMID 32333996
- [Background] Toomey D, Reid D, White S. How manual therapy provided a gateway to a biopsychosocial management approach in an adult with chronic post-surgical low back pain: a case report. J Man Manip Ther. 2021 Apr;29(2):107-132. doi: 10.1080/10669817.2020.1813472. Epub 2020 Sep 15. PMID 32930642
- [Background] Hayden JA, Ellis J, Ogilvie R, Stewart SA, Bagg MK, Stanojevic S, Yamato TP, Saragiotto BT. Some types of exercise are more effective than others in people with chronic low back pain: a network meta-analysis. J Physiother. 2021 Oct;67(4):252-262. doi: 10.1016/j.jphys.2021.09.004. Epub 2021 Sep 16. PMID 34538747
- [Derived] Vicente-Mampel J, Blanco-Gimenez P, Barrios C. Influence of patient-reported outcomes on the effect of exercise therapy, manual therapy, and kinesiotaping in chronic low back pain: secondary statistical analysis. Sci Rep. 2025 Nov 3;15(1):38400. doi: 10.1038/s41598-025-22260-3. PMID 41184444
- [Derived] Blanco-Gimenez P, Vicente-Mampel J, Gargallo P, Baraja-Vegas L, Bautista IJ, Ros-Bernal F, Barrios C. Clinical relevance of combined treatment with exercise in patients with chronic low back pain: a randomized controlled trial. Sci Rep. 2024 Jul 24;14(1):17042. doi: 10.1038/s41598-024-68192-2. PMID 39048701